CLINICAL TRIAL: NCT02273258
Title: A Randomized, Double-Blind, Controlled, Single-Dose, 3-Treatment, 3-Period, 6-Sequence Crossover Study to Compare Exposure and Activity of SAR342434 to Humalog® Using the Euglycemic Clamp Technique, in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Compare Pharmacokinetics and Pharmacodynamics of SAR342434 to Insulin Lispro in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PDY12704; 2012-004453-86; U1111-1134-4816 (Other: UTN)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — SAR342434; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (T) (Experimental): SAR342434: single dose injection
  Interventions: Drug: SAR342434
- Reference 1 (R1) (Active Comparator): US-approved Humalog®: single dose injection
  Interventions: Drug: Insulin Lispro
- Reference 2 (R2) (Active Comparator): EU-approved Humalog®: single dose injection
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: SAR342434 — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Test (T)
Drug: Insulin Lispro — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Reference 1 (R1)
Drug: Insulin Lispro — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Reference 2 (R2)

SUMMARY:
Primary Objective:

To compare exposure and activity of SAR342434 to US-approved and EU-approved Humalog®.

Secondary Objective:

To assess the safety and tolerability of SAR342434.

DETAILED DESCRIPTION:
The total study duration for a screened subject will be about 3 - 8 weeks (min-max duration, excl. screening)

* Screening: 2 to 28 days (D -28 to D -2)
* Treatment period 1 - 3: 2 days (1 overnight stay)
* Washout: 5 - 18 days (preferentially 7 days between consecutive dosing)
* End-of-study visit: 1 day between D 5 and D14 after last administration of investigational product.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects with diabetes mellitus type 1 for more than one year.
* Total insulin dose of < 1.2 U/kg/day.
* Fasting negative serum C-peptide (< 0.3 nmol/L).
* Glycohemoglobin (HbA1c) ≤ 9%.
* Stable insulin regimen for at least 2 months prior to study.
* Normal findings in medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculo-skeletal system), vital signs, electrocardiogram (ECG) and safety lab.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of insulins, thyroid hormones, lipid-lowering and antihypertensive drugs and if female with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab.
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in 1st degree relatives (parents, siblings or children).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of SAR342434, US-approved Humalog and EU-approved Humalog | 12 hours
Area under the concentration versus time curve (AUC) of SAR342434, US-approved Humalog and EU-approved Humalog | 12 hours
Area under the body weight standardized glucose infusion rate (GIR) versus time curve from 0 to 12 hours post administration (GIR-AUC0-12) | 12 hours

SECONDARY OUTCOMES:
The fractional area under the concentration versus time curve from 0 or y to x hours post administration (INS-AUC0 or Y to X) | 12 hours
Time to 20% of AUC (t20%-AUC) | 12 hours
NS-tmax, INS-t1/2z | 12 hours
The fractional area under the body weight standardized GIR versus time curve from 0 or y to x hours post administration (GIR-AUC0 or Y to X) | 12 hours
Time to 20% of total GIR-AUC0-12h (t20%-GIR-AUC0-12h) | 12 hours
Maximum smoothed body weight standardized GIR (GIRmax) | 12 hours
Time to GIRmax (GIR-tmax) | 12 hours
Duration of blood glucose control (time to elevation of smoothed blood glucose profile above clamp level and to elevation above different pre-specified blood glucose levels) | 12 hours
Number of patients with AEs, SAEs, laboratory, vital signs and electrocardiographic abnormalities , injections site reaction assessment (ISR), and if any, hypoglycemia | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi Administrative Office, Frankfurt, Germany